CLINICAL TRIAL: NCT05520645
Title: Randomized Controlled Study of Etomidate Induction in Hysteroscopic Surgery
Brief Title: Etomidate Induction in Hysteroscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 89476
Record Dates: First submitted 2022-08-19; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Etomidate Induced Dose; Hysteroscopic Surgery
MeSH Terms: interventions — Etomidate; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Eto 0.15mg/kg (Experimental): Etomidate 0.15mg/kg for anesthesia induction
  Interventions: Drug: etomidate
- Eto 0.2mg/kg (Experimental): Etomidate 0.2mg/kg for anesthesia induction
  Interventions: Drug: etomidate
- Eto 0.25mg/kg (Experimental): Etomidate 0.25mg/kg for anesthesia induction
  Interventions: Drug: etomidate
- Propofol 2mg/kg (Active Comparator): propofol 2mg/kg for anesthesia induction
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: etomidate — use etomidate for anesthesia induction in hysteroscopic surgery
  Arms: Eto 0.15mg/kg; Eto 0.25mg/kg; Eto 0.2mg/kg
Drug: propofol — use propofol for anesthesia induction in hysteroscopic surgery
  Arms: Propofol 2mg/kg

SUMMARY:
This study intends to study the optimal dose induced by etomidate in outpatients undergoing painless hysteroscopic surgery. At present, the dosage in the user manual is 0.1-0.3mg/kg. In clinical use, it is found that 0.1mg/kg often fails to achieve sedative effect, and 0.3mg/kg is prone to muscle twitching. Therefore, three groups of doses of 0.15mg/kg, 0.2mg/kg and 0.25mg/kg are set. It is hoped that this study will provide a basis for clinical evaluation of etomidate in anesthesia induction of hysteroscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients to undergo hysteroscopic surgery

Exclusion Criteria:

Hemo-dynamically unstable patients Allergic to egg protein Patients with epilepsy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-08-25 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Mean Arterial Pressure | Change in Mean Arterial Pressure(MAP) in mm of Hg from baseline value every 5 minutes for 30 minutes
  Mean value of Mean Arterial Pressures
Heart rate per minute | Change in Heart rate per minute from baseline value every five minutes for 30 minutes
  Mean of Heart rate per minute at above mentioned time intervals was measured and any study drug causing bradycardia

SECONDARY OUTCOMES:
Myoclonic movements | 60 seconds after injection of study drug
  % of cases with Myoclonic movements
Post Operative Nausea and Vomiting | Throughout entire study estimated to take 1 month to complete
  % of cases with any treatment for Post Operative Nausea and Vomiting
any oxygen saturation event below 85% by pulse oximetry | Throughout entire study estimated to take 1 month to complet
  % of cases with any oxygen saturation event below 85% by pulse oximetry

IPD SHARING:
Plan to Share IPD: No